CLINICAL TRIAL: NCT07025668
Title: Effects of Different Exercise Approaches on Tendon Cross-sectional Area and Pain in Biceps Brachii Long Head Tendinopathy
Brief Title: The Effectiveness of Different Exercise Approaches in Biceps Brachii Long Head Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Gül SEZİK, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BisepsLongHead
Record Dates: First submitted 2025-06-05; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Sports Physical Therapy; Tendinopathy
Keywords: biceps brachii; tendinopathy; tendon cross-sectional area; shoulder pain
MeSH Terms: conditions — Tendinopathy; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: three groups with a conventional therapy control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants in all three groups performed the given exercises without knowing which group they were included in. Outcome assessments will be performed by an investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Eccentric Exercise Group (Active Comparator): In the eccentric exercise group, in addition to strengthening exercises for the periscapular muscles and stretching exercises for the biceps brachii muscle, eccentric strengthening exercises for the biceps brachii muscle will be given.
  Interventions: Other: Eccentric Exercise
- Combined-Exercise Group (Active Comparator): In the combined exercise group, in addition to strengthening exercises for the periscapular muscles and stretching exercises for the biceps brachii muscle, progressive isometric, isotonic and plyometric strengthening training will be given to the biceps brachii muscle.
  Interventions: Other: Combined Exercise
- Control Group (Active Comparator): In the control group, strengthening exercises for the periscapular muscles and stretching exercises for the biceps brachii muscle will be given. Strengthening exercises for the biceps brachii muscle will not be given in this group.
  Interventions: Other: Control Group Exercise

INTERVENTIONS:
Other: Eccentric Exercise — In the eccentric exercise group, in addition to strengthening exercises for the periscapular muscles and stretching exercises for the biceps brachii muscle, eccentric strengthening exercises for the biceps brachii muscle will be given. Participants will do the exercises in the groups they were randomized to every day for 12 weeks. They will be called to the clinic once a week for exercise checks.
  Arms: Eccentric Exercise Group
Other: Combined Exercise — In the combined exercise group, in addition to strengthening exercises for the periscapular muscles and stretching exercises for the biceps brachii muscle, progressive isometric, isotonic and plyometric strengthening training will be given to the biceps brachii muscle. Participants will do the exercises in the groups they were randomized to every day for 12 weeks. They will be called to the clinic once a week for exercise checks.
  Arms: Combined-Exercise Group
Other: Control Group Exercise — In the control group, strengthening exercises for the periscapular muscles and stretching exercises for the biceps brachii muscle will be given. Strengthening exercises for the biceps brachii muscle will not be given in this group. Participants will do the exercises in the groups they were randomized to every day for 12 weeks. They will be called to the clinic once a week for exercise checks.
  Arms: Control Group

SUMMARY:
This study was planned to analyze the changes in tendon cross-sectional area and shoulder pain with different exercise approaches applied in biceps brachii long head tendinopathy.

DETAILED DESCRIPTION:
There are different conservative treatment options for biceps brachii long head tendinopathy. However, the exercise approaches that can be applied for biceps brachii tendinopathy are not clear in the literature. This study aims to investigate the effectiveness of exercises that include 12 weeks of eccentric training or combined exercise approaches.

ELIGIBILITY:
Inclusion Criteria:

* Having shoulder pain lasting 3 months or more
* Without a history of surgery, having a diagnosis of shoulder rotator cuff tendinopathy, rotator cuff stage 1-2 tear or subacromial impingement, and having been diagnosed with secondary biceps long head tendinopathy by a physician
* Pain level during activity > 3 according to the visual analog scale
* Patients who have been informed about the study and have given written consent to participate in the study will be included in the study.

Exclusion Criteria:

* Acute shoulder injury
* History of shoulder and cervical surgery
* Limitation of passive range of motion
* History of local corticosteroid injection within the last 12 months
* Patients who cannot comply with the exercise program will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Tendon Cross-Sectional Area | Baseline and 12 weeks
  Ultrasound will be used to measure tendon cross-sectional area.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline and 12 weeks
  The patient will be asked to mark the severity of his/her pain at rest, at night, and during general activity on a 10 cm line without numbers, and the point they mark will be measured in millimeters with a ruler. The left end of the line indicates no pain, corresponding to 0 cm, while the pain level increases towards the right end of the line, which is marked at 10 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru G SEZİK, Msc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman DJ, Dunn JC, Higgins LD, Warner JJ. Proximal biceps tendon: injuries and management. Sports Med Arthrosc Rev. 2008 Sep;16(3):162-9. doi: 10.1097/JSA.0b013e318184f549. PMID 18703976
- [Background] Ahrens PM, Boileau P. The long head of biceps and associated tendinopathy. J Bone Joint Surg Br. 2007 Aug;89(8):1001-9. doi: 10.1302/0301-620X.89B8.19278. PMID 17785735
- [Background] Chen RE, Voloshin I. Long Head of Biceps Injury: Treatment Options and Decision Making. Sports Med Arthrosc Rev. 2018 Sep;26(3):139-144. doi: 10.1097/JSA.0000000000000206. PMID 30059449
- [Background] Ryu JH, Pedowitz RA. Rehabilitation of biceps tendon disorders in athletes. Clin Sports Med. 2010 Apr;29(2):229-46, vii-viii. doi: 10.1016/j.csm.2009.12.003. PMID 20226316